CLINICAL TRIAL: NCT06441188
Title: Sonography of the Nipple Areolar Complex (SONAC) Study
Brief Title: Sonography of the Nipple Areolar Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christine U. Lee, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-004909
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Nipple ultrasound imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Subjects (Experimental): Healthy volunteers with no breast cancer or breast symptoms. Subjects will undergo 1 hour of non-invasive ultrasound scanning of the nipple and its adjacent tissues.
  Interventions: Diagnostic Test: Thin layer conventional ultrasound coupling gel; Diagnostic Test: Thick layer of conventional ultrasound coupling gel; Diagnostic Test: Thin conventional ultrasound coupling gel pad; Diagnostic Test: Thick conventional ultrasound coupling gel pad

INTERVENTIONS:
Diagnostic Test: Thin layer conventional ultrasound coupling gel — The GE Logiq E10 ultrasound scanner and the ML6-15 linear probe will be used to collect B-mode images of the nipple-areolar complex following routine clinical imaging practice, using a thin layer of conventional ultrasound coupling gel.
Diagnostic Test: Thick layer of conventional ultrasound coupling gel — The GE Logiq E10 ultrasound scanner and the ML6-15 linear probe will be used to collect B-mode images of the nipple-areolar complex following routine clinical imaging practice, using a thick layer of conventional ultrasound coupling gel.
Diagnostic Test: Thin conventional ultrasound coupling gel pad — The GE Logiq E10 ultrasound scanner and the ML6-15 linear probe will be used to collect B-mode images of the nipple-areolar complex following routine clinical imaging practice, using a thin conventional ultrasound coupling gel pad.
Diagnostic Test: Thick conventional ultrasound coupling gel pad — The GE Logiq E10 ultrasound scanner and the ML6-15 linear probe will be used to collect B-mode images of the nipple-areolar complex following routine clinical imaging practice, using a thick conventional ultrasound coupling gel pad.

SUMMARY:
The purpose of this study is to determine ultrasound scanning techniques of the nipple areolar complex (NAC) that provide optimal diagnostic imaging features.

ELIGIBILITY:
Inclusion Criteria:

Female, Age of 18 or older; no breast cancer; no breast symptom.

Exclusion Criteria:

Subjects lacking capacity to consent; vulnerable subjects such as prisoners.

Note: Other protocol defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Image quality satisfaction | Baseline
  Images will be ranked by three independent radiologists and scored from 1 to 4 respectively (1 is the least satisfactory, 4 is the most satisfactory).

SECONDARY OUTCOMES:
Ultrasound exam length of time | Baseline
  The total number of minutes ultrasound is performed on the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, PhD, Principal Investigator — Mayo Clinic; Shigao Chen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No